CLINICAL TRIAL: NCT01130441
Title: Study on Self-harming Behaviors of Adolescents in a Juvenile Detention House
Brief Title: Self-harming Behaviors Study of Adolescents in a Juvenile Detention House
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Mei Hua Tsai M.D., Far Eastern Memorial Hospital
Other Study IDs: 098047-3
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Adolescent Behavior; Harm Reduction
Keywords: adolescent behavior; harm reduction
MeSH Terms: conditions — Adolescent Behavior; Harm Reduction | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- self-harming group
  Interventions: Behavioral: psychotherapy
- non-self-harming group -control group

INTERVENTIONS:
Behavioral: psychotherapy — short problem-solving skills therapy intervention
  Groups: self-harming group

SUMMARY:
Incarcerated adolescents engage in suicide ideation, self-harming behaviors and have poor coping abilities, suggesting a need for mental health intervention and treatment. Previous research on self-harm among community adolescents revealed that self-harmers were more likely than non-self-harmers to report suicidal ideation, and having made a suicide plan.

This study plans to evaluate the suicidal intent of self-harming and non-self harming adolescent admitted at juvenile detention house in Taiwan. Furthermore, this study also plans to identify the prevalence and types of self-harming activities of incarcerated youths. Another purpose is to investigate the coping abilities of incarcerated youth, with evaluation of efficacy of short problem-solving skills therapy intervention by trained psychologists of three sessions for adolescents with poor coping adjustment; referral to adolescent psychiatrist when severe mental disorder or poor coping abilities were found.

By analyzing their suicidal ideation, self-harming behaviors, and coping adjustment, the investigators will be able to give timely intervention and identify effective means and methods for better serving this population. This study hopes to help the incarcerated youth to replace their self-destructive behaviors with effective coping adjustment abilities.

DETAILED DESCRIPTION:
Suicide among youth ranked third in Taiwan. According to a study by Lin, stressors include family, school and friends. Psychiatric symptoms also played a role (Lin, 2002) . Incarcerated adolescents with poor coping adjustment will be referred to psychologists. The psychologists were trained by the juvenile detention adolescent psychiatrist.

Taiwanese adolescents have very high rate of self-harming activities, furthermore, incarcerated adolescents are expected to have a higher rate of self-harming activities. There are few studies done on self-harming activities, suicidal intent and coping style of incarcerated youth in Taiwan. According to a study on self-harming adolescents in a juvenile correctional facility, these youth have higher rates of suicide attempts and use more violent methods of attempt than adolescents in the general population (Penn, 2003). They also have poor problem-solving skills. We hope to study their suicidal ideations, self-harming behaviors, and coping styles in order to offer appropriate and timely intervention. We can then offer skills to deal with similar triggering events in the future.

Furthermore, it is hoped that recidivism can be reduced after psychopathological intervention.

ELIGIBILITY:
Inclusion Criteria:

* youth admitted at juvenile detention center on Jan 1,2010 up to Dec 31,2010

Exclusion Criteria:

* currently emotionally unstable, are suffering from active psychotic process like schizophrenia, mentally retarded, illiterate or refuse to participate.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Youth admitted at juvenile detention center in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei Hua Tsai, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Juvenile Detention Center Taipei, Taipei, Taipei Hsian, Taiwan